CLINICAL TRIAL: NCT00946036
Title: Bioequivalence Study of Sertraline 100 mg Tablet and ZOLOFT Following a 100 mg Dose in Healthy Subjects Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: 40486
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
MeSH Terms: interventions — Sertraline

INTERVENTIONS:
Drug: Sertraline Hydrochloride

SUMMARY:
* Objective:

  * To compare the rate and extent of absorption of Torrent Pharmaceuticals Limited, India, sertraline and Pfizer, Inc., USA (Zoloft) sertaline, administered as a 1X100 mg tablet, under fasted conditions.
* Study Design:

  * Single-dose, open-label, randomized two-way crossover.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, smoker or non smoker, 18 years of age and older.
* Capable of consent.
* BMI>= 19.0 and <30.0 kg/m2

Exclusion Criteria:

* Clinically significant illness or surgery within 4 weeks prior to the administration of the study medication.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities or vital sign abnormalities(blood pressure).
* History of significant alcohol or drug abuse within one year prior to the screening visit.
* History or allergic reactions to heparin, sertraline or other related drugs.
* Use of an investigational drug or participation in an investigational study with in 30 days prior to administration of the study medication.
* Clinically significant history of gastrointestinal pathology, liver or kidney disease, neurological, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* History of seizures, suicide attempt, bipolar disorder or manic episodes.
* Depot injection or an implant of any drugs with in 6 months prior to administration of study medication.
* Breastfeeding subject.
* Positive urine pregnancy test at screening.
* Female subject of child bearing potential having unprotected sexual intercourse with any non-sterile mail partner within 14 days prior to study drug administration. Acceptable methods of contraception:

  1. Intra-uterine contraceptive device(placed at least 4 weeks prior to study drug administration)
  2. Condom or diaphragm + spermicide.

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Anapharm Inc., Montreal, Quebec, Canada